CLINICAL TRIAL: NCT03160495
Title: Functional ImaGing of Heterogeneity in Head and Neck Tumors - Validation From Surgical Specimens
Acronym: FIGHHT
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jacob Rasmussen, MD, PhD, Rigshospitalet, Denmark
Other Study IDs: H-16049387
Record Dates: First submitted 2017-05-16; First posted 2017-05-19 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: PET/MR; Squamous cell carcinoma; Heterogeneity
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — The gross specimen will be examined, sectioned and placed in tissue cassettes as done in routine. Six tissue blocks will be picked for microscopic evaluation and IHC staining. The specific selection of cancer related IHC biomarkers is based on their relationship with tumor cell metabolism, radiotherapy resistance (proliferation and hypoxia), association with FDG accumulation and institutional experience from a previous study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: All patients — All patients are scanned with PET/MR prior to surgery.

SUMMARY:
The purpose of this study is to investigate if heterogeneity in head and neck squamous cell carcinoma as seen in functional imaging with PET/MR can be correlated to biologic heterogeneity in surgical specimens.

DETAILED DESCRIPTION:
The following is a presentation of a prospective protocol, named FIGHHT, including patients with squamous cell carcinoma of the head and neck (HNSCC) who are referred for surgery.

This is a prospective imaging/biomarker expression study where patients referred for surgery for HNSCC will be included. The purpose of the study is to investigate if heterogeneity in HNSCC as seen in functional imaging with PET/MR can be correlated to biologic heterogeneity in surgical specimens.

Multiparametric imaging(MPI) is performed before surgery using a PET/MR system (Siemens Biograph mMR) with a 3 T magnet using a head and neck coil. The scan protocol includes diffusion weighted MRI, dynamic contrast enhanced perfusion MRI and FDG-PET (4 MBq/kg). Morphometric imaging is performed with a 3D T2 weighted sequence (SPACE, voxel size 1.0 mm isotropic in vivo and 0.5 mm isotropic for specimens).

The scans are evaluated by a radiologist and a specialist in nuclear medicine and regions of interest and reference areas (anatomical landmarks) are marked. The tumor and if indicated lymp nodes are removed en bloc and per-operatively the reference areas and other anatomical landmarks are marked in the specimen with intravenous tubes. The specimen is fixed to a corkboard and scanned morphometric (as described) using a knee coil before and after formalin fixation within 1 hour after surgery. The whole surgical specimen is sectioned for histological processing.

Tissue blocks will undergo microscopic pathological evaluation and IHC staining. The specific selection of cancer related IHC biomarkers is based on their relationship with tumor cell metabolism, radiotherapy resistance (proliferation and hypoxia), association with FDG accumulation and institutional experience from a previous study.

The quantified measurements from the FDG PET, DWI and DCE scan will be correlated to the expression of IHC biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age above 18
* Primary or recurrent squamous cell carcinoma in the head and neck area
* Referred to surgery
* Primary tumor > 1.5 cm and or neck metastasis of more than 1 cm.

Exclusion Criteria:

* Patient refusal
* Contraindications for FDG-PET/MR scan

  * Pacemaker
  * Severe claustrophobia
  * Magnetic metal in the body that is not MR compatible

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Please see detailed description
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Quantified measures from FDG PET and pathology | 3-6 months
  Correlation between FDG uptake (measured as SUV) and expression of IHC biomarkers
Quantified measures from DWI and pathology | 3-6 months
  Correlation between diffusion weighted imaging and expression of IHC biomarkers
Quantified measures from DCE and pathology | 3-6 months
  Correlation between dynamic contrast enhancement and expression of IHC biomarkers

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Otorhinolaryngology, Head & Neck Surgery and Audiology Rigshospitalet, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No